CLINICAL TRIAL: NCT00694876
Title: Impact of Health Literacy and Other Factors on Glaucoma Patient Adherence in South India
Status: Completed | Type: Observational
Sponsor: Robin, Alan L., M.D. (Individual)
Responsible Party: Sponsor
Other Study IDs: Health Literacy
Record Dates: First submitted 2008-06-07; First posted 2008-06-11 (Estimated); Last update posted 2012-11-30 (Estimated); Status verified 2012-11

CONDITIONS: Patient Noncompliance; Health Literacy; Glaucoma
Keywords: Health Literacy; Patient Nonadherence; Patient Noncompliance; Follow Up; India; Glaucoma
MeSH Terms: conditions — Patient Compliance; Glaucoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Adequate Health Literacy (as determined by TOFHLA)
- 2: Inadequate Health Literacy (as determined by TOFHLA)

SUMMARY:
The purpose of this study is to determine how health literacy impacts glaucoma patient adherence (as measured by following up with the doctor) in Tamil Nadu, India. We hypothesize that individuals with better health literacy will have higher rates of follow-up with their ophthalmologist.

DETAILED DESCRIPTION:
Many studies have shown the importance of health literacy on patient adherence in the United States (Juzych, M, et al., 2008; Muir, KW, et al., 2006). Low adherence in glaucoma patients leads to increased intraocular pressure, optic nerve damage, and blindness. To date, no research has been done with health literacy and patient adherence in the developing world.

We will use TOFHLA and REALM to assess the health literacy of glaucoma patients in Tamil Nadu, India. We will also survey other demographic information and patient knowledge of glaucoma. This information will be compared with follow-up rates to identify barriers to patient adherence.

ELIGIBILITY:
Inclusion Criteria:

* Better than 20/100 corrected vision in better eye
* Must live within 50 miles of Aravind Eye Hospital
* Clinical diagnosis of primary glaucoma
* Paying patient

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Glaucoma Patients from Aravind Eye Hospital at Madurai, Tamil Nadu, India
Sampling Method: Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2008-06; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Association between TOFHLA and REALM and the probability of return for follow-up visit | 1 year from enrollemnt

SECONDARY OUTCOMES:
Association between religion, caste, education, socio-economic status, employment, and available time for doctor visits and the probability of return for follow-up visit. | 1 year from enrollment
Association between marital status, number of dependents, family history of glaucoma, travel, need for an escort, understanding of glaucoma, and paying status and the probability of return for follow-up visit. | 1 year from enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin R Curran, BS, Principal Investigator — Loyola University Chicago, Stritch School of Medicine; Alan L Robin, MD, Study Director — University of Maryland; Johns Hopkins University, Wilmer Institute and Bloomberg School of Public Health; Ramaswami Krishnadas, DO, DNB, Study Director — Aravind Eye Hospital, CMO; Scott D Smith, MD, MPH, Study Director — The Cleveland Clinic
Locations (1):
- Aravind Eye Hospital, Madurai, Tamil Nadu, India

REFERENCES:
- [Background] Juzych MS, Randhawa S, Shukairy A, Kaushal P, Gupta A, Shalauta N. Functional health literacy in patients with glaucoma in urban settings. Arch Ophthalmol. 2008 May;126(5):718-24. doi: 10.1001/archopht.126.5.718. PMID 18474786
- [Background] Muir KW, Santiago-Turla C, Stinnett SS, Herndon LW, Allingham RR, Challa P, Lee PP. Health literacy and adherence to glaucoma therapy. Am J Ophthalmol. 2006 Aug;142(2):223-6. doi: 10.1016/j.ajo.2006.03.018. PMID 16876500
- [Background] Friedman DS, Hahn SR, Gelb L, Tan J, Shah SN, Kim EE, Zimmerman TJ, Quigley HA. Doctor-patient communication, health-related beliefs, and adherence in glaucoma results from the Glaucoma Adherence and Persistency Study. Ophthalmology. 2008 Aug;115(8):1320-7, 1327.e1-3. doi: 10.1016/j.ophtha.2007.11.023. Epub 2008 Mar 5. PMID 18321582